CLINICAL TRIAL: NCT01714167
Title: Autologous Bone Marrow Mesenchymal Stem Cell Transplantation for Treatment of Chronic Stroke
Brief Title: Autologous Bone Marrow Mesenchymal Stem Cell Transplantation for Chronic Stroke
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wenzhou Medical University (Other)
Collaborators: University of North Texas Health Science Center (Other)
Responsible Party: Principal Investigator, Qichuan Zhuge, Department of Neurosurgery, Wenzhou Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WZMC-2011-8
Record Dates: First submitted 2012-10-19; First posted 2012-10-25 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Stroke
Keywords: Chronic; Ischemic Stroke; Intracerebral Hemorrhage; Bone Marrow Mesenchymal Stem Cell
MeSH Terms: conditions — Stroke; Bronchiolitis Obliterans Syndrome; Ischemic Stroke; Cerebral Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- intracerebral stem cell transplantation (Active Comparator): Intracerebral transplantation of autologous bone marrow mesenchymal stem cell, 2-4 million stem cells per patient plus conventional treatment include rehabilitation
  Interventions: Genetic: intracerebral stem cell transplantation
- conventional treatment (No Intervention): Control group receive conventional stroke treatment that include rehabilitation

INTERVENTIONS:
Genetic: intracerebral stem cell transplantation — Intracerebral transplantation of autologous bone marrow mesenchymal stem cell, 2-4 million stem cells per patient
  Arms: intracerebral stem cell transplantation

SUMMARY:
Stroke is one of the leading causes of disability in the world, and stem cell - transplantation provides a promising approach for rehabilitation. The main objective of this study is to evaluate the efficacy of the intracerebral injection of autologous bone marrow mesenchymal stem cells in patients with chronic stroke.

DETAILED DESCRIPTION:
For many stroke survivors, the best hope is a lengthy program of rehabilitation, followed by a life-long process of clinical support. However, even with rehabilitation therapy, 50% to 95% of stroke survivors remain impaired. There is thus a great need for new therapeutic developments for patients with disability after stroke, which is largely unexplored. Regenerative cell-based therapies offer long-term hope for many patients with stroke, as stem cells might be possible for dead or injured neural cells to be replaced after acute stroke. In this study, the investigators will assess the safety and feasibility of intracerebral transplantation of autologous bone marrow mesenchymal stem cells in patients with chronic stroke. The neurological outcome will be determined after transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Aged 40-70 ischemia stroke or intracerebral hemorrhage patient
* With stroke history of more than 3 months, less than 60 months
* With stable hemiplegia condition
* NIHSS (NIH stroke scale) score of 7 or more points
* Patient is stable (normal respiration, afebrile, BP less than mean arterial pressure of 125 mm of Hg, fasting blood sugar <7 mg, and normal urea/electrolytes for at least 48 hours.)

Exclusion Criteria:

* Patients aged less than 40 or more than 70
* Lacunar infarction
* History of neurological disease, head injury or psychiatric disorder with disablity
* Pregnant women
* Impaired liver function, abnormal blood coagulation, AIDS, HIV, combine other tumor or special condition
* Inaccessibility for follow up
* Unwillingness to provide written informed consent

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-06; Primary Completion 2015-10 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in NIH Stroke Scale at 12 months | 1, 6 and 12 months

SECONDARY OUTCOMES:
Improvement of infarct size measured by brain MRI | 1,6 and 12 months after transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Kunlin Jin, M.D., Ph.D., Study Director — University of North Texas Health Science Center; Qichuan Zhuge, M.D., Study Chair — First Affiliated Hospital of Wenzhou Medical University
Locations (1):
- The First Affiliated Hospital of Wenzhou Medical College, Wenzhou, Zhejiang, China